CLINICAL TRIAL: NCT04706221
Title: Clinical Evaluation of the CM-1500 in Postoperative Abdominal and Pelvic Surgery Patients
Brief Title: Clinical Evaluation of the CM-1500 in Postoperative Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Monitoring Solutions (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZMS-1500-2001
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single-arm, non-randomized, non-controlled, single-center study enrolling adult subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Blood Volume Monitoring (Experimental)
  Interventions: Device: CM-1500

INTERVENTIONS:
Device: CM-1500 — Blood volume monitor CM-1500

SUMMARY:
The primary objective is to evaluate the the changes in the Relative Index in post abdominal or pelvic surgery patients on the Cardiac Monitor Model CM-1500.

DETAILED DESCRIPTION:
Postoperative hemorrhage incidence can vary depending on the type of surgery, but it can lead to severe clinical complications ranging from mild anemia to fatal hemorrhagic shock. Monitoring and detecting these fluid changes postoperatively can be complicated, and standard operating procedures vary. The Cardiac Monitor, Model 1500 (CM-1500), uses a personalized approach by non-invasively and simultaneously monitoring five (5) physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Ability and willingness to comply with study procedures and duration requirements
* 18 years of age or older
* Undergoing an abdominal or pelvic surgery within the next 10 days

Exclusion Criteria:

* Females who are pregnant or breastfeeding
* Participation in other clinical studies involving experimental drugs or devices
* Undergone an amputation of the left upper extremity
* Diagnosed with Dextrocardia
* Subjects who have a Pacemaker

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Volume Monitoring - Open Surgery: Monitoring with CM-1500 (Blood volume monitor CM-1500) during Open Surgery
- Blood Volume Monitoring - Laparoscopic Surgery: Monitoring with CM-1500 (Blood volume monitor CM-1500) during Laparoscopic Surgery
Period: Overall Study
Arm/Group | Blood Volume Monitoring - Open Surgery | Blood Volume Monitoring - Laparoscopic Surgery
Started | 91 | 109
Completed | 75 | 98
Not Completed | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Blood Volume Monitoring Laparoscopic Surgery: CM-1500: Blood volume monitor post-laparoscopic surgery
- Blood Volume Monitoring - Open Surgery: CM-1500: Blood volume monitor post-open surgery
- Total: Total of all reporting groups
Arm/Group | Blood Volume Monitoring Laparoscopic Surgery | Blood Volume Monitoring - Open Surgery | Total
Number analyzed (Participants) | 98 | 75 | 173
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 70 | 45 | 115
  >=65 years | 28 | 30 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (14.3) | 58.4 (15.2) | 56.25 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 40 | 102
  Male | 36 | 35 | 71
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 98 | 75 | 173

OUTCOME MEASURES:

1. Primary Outcome: Relative Index Change During PACU Stay
Description: The primary objective is to evaluate changes in the Relative Index (RI) in post-abdominal or pelvic surgery patients (Laparoscopic or Open). The CM-1500 monitors parameters which are indicative of relative changes in fluid volume in adult patients. The Relative Index is an investigational value which utilizes proprietary algorithms to combine the relative changes of each measured parameter into a single value. The Relative Index is graded on a scale where 100 indicates a patient's baseline, and changes up or down from the baseline could be used as potential indicators of fluid gain or loss relative to the baseline, based on the changes of the individually monitored parameters. Per the device's FDA 510(k) clearance, the RI is computed as the weighted summation of the percent change values (signifying the deviation of each parameter from it's baseline value) for its parameters. Change in RI is calculated by subtracting the initial RI value from the final RI value during monitoring.
Time Frame: Length of PACU Stay (Range: 46 to 353 minutes)
Measure: Mean (Standard Deviation); unit: Relative Index (RI)
Groups:
- Blood Volume Monitoring - Open Surgery: CM-1500: Monitoring with CM-1500 (Blood Volume Monitor CM-1500) during Open Surgery
- Blood Volume Monitoring - Laparoscopic Surgery: CM-1500: Monitoring with CM-1500 (Blood Volume Monitor CM-1500) during Laparoscopic Surgery
Arm/Group | Blood Volume Monitoring - Open Surgery | Blood Volume Monitoring - Laparoscopic Surgery
Number analyzed (Participants) | 75 | 98
Relative Index (RI) | -2.01 (4.00) | -1.32 (3.11)

ADVERSE EVENTS:
Time Frame: Subject adverse event data were collected while patients were in PACU (range: 46 - 353 minutes).
Arm/Group | Blood Volume Monitoring Laparoscopic Surgery | Blood Volume Monitoring - Open Surgery
All-Cause Mortality (participants affected / at risk) | 0/98 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/98 | 0/75
Other Adverse Events (participants affected / at risk) | 0/98 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/21/NCT04706221/Prot_SAP_000.pdf